CLINICAL TRIAL: NCT01702922
Title: Understanding the Perceived Influence of Childhood Cancer and NF1 on the Parents' Marital/Partner Relationship: A Descriptive Study
Brief Title: Relationship Stressors in Parents of Children With Cancer or Neurofibromatosis Type 1 (NF1)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120206; 12-C-0206
Record Dates: First submitted 2012-10-06; First posted 2012-10-10 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Parents of Children With Cancer; Parents of Children With NF1; Parents of Children With Neurofibromatosis Type I
Keywords: Stress; Marriage; Dyadic Coping; Mother; Father; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1/Active Cancer Parents: Must have been in a partnership at the time child was diagnosed with cancer & must have been diagnosed at least 3 months prior to enrollment on this study & be currently receiving treatment
- 2/Complete Cancer Parents: Must have been in a partnership at the time the child was diagnosed with cancer and the child has completed treatment at age 21 or younger (without evidence of disease) within the previous 3 years
- 3/NF1 Parents: Must have been in a partnership at the time the child was diagnosed with NF1 and the child must have been diagnosed with NF1 at least 3 months prior to enrollment on this study.

SUMMARY:
Background:

- Serious illnesses like cancer or Neurofibromatosis Type 1 (NF1), can cause high levels of stress in a family. When a child is diagnosed with cancer or NF1, parents face numerous stressors, each of which can strain relationships. Many parents struggle to effectively cope with the changes in parenting roles that often accompany treatment of childhood cancer or NF1. How parents cope with this stress can influence whether the relationship is strengthened or weakened. Stress levels can also affect the care of the child who has cancer or NF1. Researchers want to better understand the critical time points and events during the child s treatment when the relationship becomes most stressed and/or strengthened.

Objectives:

- To study how stress affects the relationship between parents who have a child with cancer or Neurofibromatosis Type 1 (NF1).

Eligibility:

* Parents of a child (between 1 and 24 years of age) who has been diagnosed with cancer or NF1.
* Participants must have been in a partnership at the time the child was diagnosed with cancer or NF1. At least one of the parents must be a biological or legal parent of the child.

Design:

* Participants will fill out a questionnaire either online or by paper and pencil. It will take about 20 minutes to complete. The questions ask about the experience of dealing with a child s cancer OR NF1 diagnosis and how it affects participants relationship with their spouse/partner.
* Some participants will also have an in-depth interview. It will last about an hour. It will ask further questions about the cancer OR NF1 diagnosis and treatment and its effect on the relationship.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Background:

* Parents face numerous stressors when their child is diagnosed with cancer or NF1, each of which can strain a marriage/partnership.
* Marital/partner relationship dynamics are often not assessed or addressed when providing health care for children with cancer or NF1. Many parents struggle to effectively cope with the changes in parenting roles that frequently accompany treatment of childhood cancer or NF1.
* How parents cope with these stressors can strengthen or weaken the relationship, and can impact the entire family, including the care to the child undergoing cancer or NF1 treatments.
* Limited studies have examined relationship stress or satisfaction during a child s illness trajectory for cancer or NF1 or the critical time points and events during the child s illness trajectory when the relationship becomes most stressed and/or strengthened.

Objectives:

* To explore whether the stress associated with having a child with cancer or NF1 is perceived to impact the communication between partners.
* To explore whether positive dyadic coping (joint decision making, joint problem solving, sharing responsibilities) is perceived to have strengthened the marital relationship/partnership following the child s diagnosis with cancer or NF1.
* To describe the time points and events during the child s illness trajectory when the parents relationship becomes most stressed and/or strengthened.
* To compare the perceptions of various subgroups in the sample, (e.g. parents who score either high or low on a marital stress scale, mothers versus fathers) statistically or qualitatively as the distribution of the characteristics of the sample allow.

Eligibility:

* Participants must have been in a partnership at the time the child was diagnosed with cancer or NF1. At least one of the participating parents must be a biological or legal parent of the child. If a divorce/separation occurred with a previous partner during/after the child s diagnosis, the other partner will be invited to participate.
* The participant s child must be between 1-24 years of age.
* There are 3 groups of participants being recruited: 1) those who have a child who has been diagnosed with cancer at least 3 months prior to enrolling on this study and are currently undergoing cancer treatment, 2) those who have completed treatment at age 21 or younger (without evidence of disease) within the previous 3 years, and 3) those who have a child who has been diagnosed with NF1 at least 3 months prior to enrolling on this study.
* Participants must be fluent in the English language
* The participant s child must have been diagnosed with cancer or NF1 at least 3 months prior to enrollment on this study.
* Participants must verbalize willingness to discuss the impact of their child s cancer or NF1 diagnosis on their relationship.

Design:

* Cross-sectional, multi-center, exploratory study utilizing a convenience sample to explore the parents perception of how the child s cancer or NF1 diagnosis, treatment, decision making and other aspects of care are addressed and impact the martial relationship/partnership.
* Subjects will complete a self-administered measure that addresses potential stresses experienced in the partnership since the child s diagnosis and how each are either resolved or create a divide in the relationship.
* Subjects who experience a high or low degree of relationship stress on a standardized marital stress form (a score greater than one standard deviation from the norm) will be invited to participate in a qualitative interview, that further explores which components of parenting a child with cancer is most challenging on the relationship.
* Up to 360 participants will be enrolled onto this study (up to 180 couples). Subjects may be offered a gift card ($20 Target gift card at NIH) upon completion of the questionnaire for their time and inconvenience, where available. Due to limitations with funding, participants enrolled after July 2016 will not receive a gift card.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have been in a partnership at the time the child was diagnosed with cancer or NF1. At least one participant must be the biological/legal parent of the child; the partner may or may not be a biological/legal parent. Divorced parents who separated or divorced during or after the child s treatment can participate in this study.
* The participant s child must be between 1-24 years of age.
* Participants must be 18 years of age or older.
* Participants must be fluent in the English language.
* The participant s child must have been:

  * diagnosed with cancer at least 3 months prior to enrollment on this study and be currently receiving treatment OR
  * have completed treatment at age 21 or younger (without evidence of disease) within the previous 3 years OR
  * diagnosed with NF1 at least 3 months prior to enrollment on this study
* Participants must verbalize willingness to discuss the impact of their child s cancer or NF1 diagnosis on their relationship.
* Able to understand and willing to sign the informed consent document.

EXCLUSION CRITERIA:

* Parents of a child with cancer OR NF1 without a partner/spouse during the child s treatment for cancer or NF1 are excluded from this study.
* Parents who were not living with the child during his or her treatment and involved in the child s care.
* Parents of children who are enrolled in hospice care.
* Presence of psychotic symptoms or severe psychological distress, which in the judgment of the Principal or Associate Investigator would compromise the participants ability to engage in the study procedures or results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have been in a partnership at the time the child was diagnosed with cancer or NFl. At least one participant must be the biological/legal parent of the child; the partner may or may not be a biological/legal parent. Divorced parents who separated or divorced during or after the child's treatment can participate in this study.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Stress impact communication | 3 months
  To explore whether the stress associated with having a child with cancer or NF1 is perceived to impact the communication between partners.

SECONDARY OUTCOMES:
Dyadic coping | 3 months
  To explore whether positive dyadic coping (joint decision making, joint problem solving, sharing responsibilities) is perceived to have strengthened the marital relationship/partnership since the child s diagnosis with cancer or NF1.
Stressful timepoints | 3 months
  To describe the time points and events during the child s illness trajectory when the relationship becomes most stressed and/or strengthened.
Perception comparison | 3 months
  To compare the perceptions of various subgroups in the sample, (e.g. parents who score either high or low on a marital stress scale, mothers versus fathers) statistically or qualitatively as the distribution of the characteristics of the sample allow.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Wiener, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
- Alberta's Children's Hospital Hematology/Oncology/Transplant Program, Alberta, Canada

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0206.html